CLINICAL TRIAL: NCT01259869
Title: A Phase II Study of PX-866 in Patients With Glioblastoma Multiforme at Time of First Relapse or Progression
Brief Title: A Study of PX-866 in Patients With Glioblastoma Multiforme at Time of First Relapse or Progression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Cascadian Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I204
Record Dates: First submitted 2010-12-09; First posted 2010-12-14 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2020-05

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — PX-866

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PX-866 (Experimental)
  Interventions: Drug: PX-866

INTERVENTIONS:
Drug: PX-866 — 1 cycle = 8 weeks on study PX-866 - 8mg PO Daily

SUMMARY:
The purpose of this study is to find out whether the new drug PX-866 will slow the growth of your glioblastoma multiforme.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of glioblastoma multiforme (GBM), with recurrent or progressive disease following or during primary treatment not curable with standard therapies.
* All patients must have formalin fixed paraffin embedded tissue available for translational studies.
* Presence of bidimensionally measurable enhancing lesions on CT or MRI, with at least one lesion with a minimum dimension of 1 cm x 1 cm (i.e. both dimensions must be ≥ 1.0 cm). Baseline CT or MRI must be done within 14 days prior to registration.
* ECOG performance of 0, 1 or 2.
* Age ≥ 18 years of age. Previous Therapy

Chemotherapy:

Patients may have received prior adjuvant chemotherapy and/or concurrent chemoradiation as part of primary therapy, but must have received no therapy for recurrent/ progressive GBM (i.e. PX-866 must be first treatment for recurrence/ progression). A minimum of 28 days since the last dose of chemotherapy must have elapsed prior to registration.

Targeted Therapy:

No prior therapy with a phosphatidylinositol 3-kinase (PI-3K) inhibitor. Other targeted agents are permissible provided they were given as part of front line treatment. A minimum of 56 days (8 weeks) must have elapsed since last day for anti-angiogenic therapy and minimum of 28 days for other targeted agents.

Radiation:

Patients may have had prior radiation therapy provided at least 28 days have elapsed from the day of the last fraction of radiation to the date of registration.

- Previous Surgery: Previous surgery is permitted provided that wound healing has occurred and at least 14 days have elapsed prior to registration.

5.1.7 Laboratory Requirements (must be done within 7 days prior to registration)

Hematology:

Granulocytes (AGC) ≥ 1.5 x 109/L Platelets ≥ 100 x 109/L

Chemistry:

Serum creatinine ≤ 1.5 x UNL Total bilirubin ≤ 1.5 x UNL ALT and AST ≤ 1.5 x UNL Glucose ≤ 8.9 mmol/L (≤ Grade 1)

* Women must be post menopausal, surgically sterile or use a reliable form of contraception while on study and for 30 days after discontinuing therapy. Women of childbearing potential must have a pregnancy test taken and proven negative within 7 days prior to registration and must not be lactating.
* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements. It will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the NCIC CTG Study Coordinator that such clearance has been obtained, before the trial can commence in that centre. Because of differing requirements, a standard consent form for the trial will not be provided but a sample form is provided. A copy of the initial full board REB approval and approved consent form must be sent to the central office. The patient must sign the consent form prior to registration (exception for translations). Please note that the consent form for this study must contain a statement which gives permission for the NCIC CTG and monitoring agencies to review patient records Patients who cannot give informed consent (i.e. mentally incompetent patients, or those physically incapacitated such as comatose patients) are not to be recruited into the study. Patients competent but physically unable to sign the consent form may have the document signed by their nearest relative or legal guardian. Each patient will be provided with a full explanation of the study before consent is requested.
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 2 hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves that the patients registered on this trial will be available for complete documentation of the treatment, adverse events, response assessment and follow-up.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 2 working days of patient registration.

Exclusion Criteria:

* Patients who have other active malignancies (i.e. documented by imaging, clinical exam or marker) are to be excluded. (Please call NCIC CTG if any questions about the interpretation of this criterion).
* Known HIV-positive patients.
* Uncontrolled diabetes mellitus.
* Patients should be on a stable dose of steroid (i.e. no change in dose for 2 weeks prior to registration) when entered on study. Patients recently started on steroids or whose steroid dose was increased in the recent past should not be started on protocol treatment until at least 2 weeks have passed from the time of steroid dose increment or initiation. Under these circumstances, baseline CT or MRI scan for purposes of assessment of response to protocol treatment should be done at the time of initiation of protocol therapy (i.e., these patients must be re-imaged to control for steroid effects).

Note:

The idea behind this is to restrict entry to a subset of patients who are not rapidly changing: especially rapidly deteriorating. If a patient being worked up for the trial appears to need to have steroid introduced or increased, the patient should be treated as is medically appropriate (i.e., have the steroid introduced or increased). Steroid should NOT be withheld if clinically indicated just so that patients can be registered on study!

* Patients with upper gastrointestinal or other conditions that would preclude compliance or absorption of oral medication are not eligible.
* Patients with active or uncontrolled infections, or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol.
* Patients are not eligible if they have a known hypersensitivity to the study drugs or their components.
* Patients who have had prior treatment with a PI3 kinase inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2014-10-29 (Actual); Study Completion 2015-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Pitz, Study Chair — CancerCare Manitoba
Locations (7):
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - London Regional Cancer Program, London, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pitz MW, Eisenhauer EA, MacNeil MV, Thiessen B, Easaw JC, Macdonald DR, Eisenstat DD, Kakumanu AS, Salim M, Chalchal H, Squire J, Tsao MS, Kamel-Reid S, Banerji S, Tu D, Powers J, Hausman DF, Mason WP. Phase II study of PX-866 in recurrent glioblastoma. Neuro Oncol. 2015 Sep;17(9):1270-4. doi: 10.1093/neuonc/nou365. Epub 2015 Jan 20. PMID 25605819

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PX-866
Started | 34
Completed | 33
Not Completed | 1
Not completed — Duplicated registration | 1

BASELINE CHARACTERISTICS:
Population: All patients completed the study
Arm/Group | PX-866
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 56 [35 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 33

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Assessed by evaluation of change in product of bidimensional measurement of enhancing brain tumour on CT scan or MRI
Time Frame: 18 months
Population: All patients completed study
Measure: Count of Participants; unit: Participants
Arm/Group | PX-866
Number analyzed (Participants) | 33
Participants | 1

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | PX-866
All-Cause Mortality (participants affected / at risk) | 15/33
Serious Adverse Events (participants affected / at risk) | 9/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PX-866 (N=33)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increase (Investigations) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Seizure (Nervous system disorders) | 3 (3)
Eye pain (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Death NOS (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PX-866 (N=33)
Hearing impaired (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Cushingoid (Endocrine disorders) | 2
Blurred vision (Eye disorders) | 5
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 7
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 15
Death NOS (General disorders) | 2
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 23
Gait disturbance (General disorders) | 2
Urinary tract infection (Hepatobiliary disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Ataxia (Nervous system disorders) | 3
Concentration impairment (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 3
Dysarthria (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Dysphasia (Nervous system disorders) | 9
Facial nerve disorder (Nervous system disorders) | 3
Headache (Nervous system disorders) | 21
Memory impairment (Nervous system disorders) | 4
Peripheral motor neuropathy (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 3
Pyramidal tract syndrome (Nervous system disorders) | 6
Seizure (Nervous system disorders) | 11
Tremor (Nervous system disorders) | 2
Other nervous system disorders (Nervous system disorders) | 6
Anxiety (Psychiatric disorders) | 7
Confusion (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 10
Urinary frequency (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 3
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No